CLINICAL TRIAL: NCT06165705
Title: Treating Amblyopia With CureSight
Acronym: ABCDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABCD CureSight
Record Dates: First submitted 2023-12-04; First posted 2023-12-11 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-01

CONDITIONS: Amblyopia
Keywords: refractive amblyopia, strabismic amblyopia, anisometropia
MeSH Terms: conditions — Amblyopia; Anisometropia | interventions — Eye-Tracking Technology

STUDY DESIGN:
Intervention Model Description: treatment efficacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Amblyopia therapy with Curesight outside FDA limited ranges (Experimental): Severity of amblyopia and age range outside FDA study
  Interventions: Device: CureSight

INTERVENTIONS:
Device: CureSight — dichoptic therapy with anaglyph goggles and eye tracking
  Other Names: dichoptic therapy with anaglyph goggles and eye tracking

SUMMARY:
Patients with visual acuity and ocular characteristics outside the Novasight FDA multi-center study are to perform the same Curesight procedures- including M&S EVA or eETDRS patched acuity, stereo and then utilize the Curesight device 1.5 hours per day, 6 days per week over 3-6 months to determine treatment efficacy.

An Eye-Tracking-Based Dichoptic Home Treatment for Amblyopia: A Multicenter Randomized Clinical Trial T. Wygnanski-Jaffe, B. J. Kushner, A. Moshkovitz, M. Belkin, O. Yehezkel and G. CureSight Pivotal Trial Ophthalmology 2023 Vol. 130 Issue 3 Pages 274-285

DETAILED DESCRIPTION:
Patients with visual acuity worse than 20/30 due to amblyopia will be offered therapy with Curesight. The Curesight-component of amblyopia therapy will be offered no-charge for up to 4 months. The Curesight device must then be returned to Alaska Blind Child Discovery.

The Curesight device will be administered in a similar, safe manner as the previous multi-centered trial that was performed in Israel and the US.

Patient Selection Inclusion criteria: patients aged 3 to less than 19 years. Amblyopia may be due to refractive error, strabismus and/or deprivation.

Exclusion criteria: Inability to participate with any form of monocular visual acuity testing and stereopsis testing. Light-induced seizures. Lack of any internet at home. Pregnancy.

Recruitment: Patients will be recruited from within Alaska Children's EYE & Strabismus clinical practice. Patients will not be paid for recruitment. Patients will have opportunity to review the publication regarding the study1.

Protocol (from Curesight Pivotal Trial NS-00706-R01) Binocular CureSight Treatment CureSight™ is an eye-tracking-based, dichoptic system aimed for the treatment of amblyopia under dichoptic conditions. The technology is based on real-time eye tracking and separation of the visual stimuli presented on a monitor into two separate digital channels, one for each eye. Using this dichoptic method, any online content can be tailored individually per eye and then presented simultaneously to each eye. During the treatment, dichoptic anaglyph glasses that are part of the CureSight™ system have to be worn over the habitual spectacle correction. In short, the technology has 2 main components: 1. Eye-tracker and anaglyph glasses that allow continuous gaze position tracking for each eye and image presentation in the optimum position to each eye, including cases of eye deviation and 2. Software that blurs the non-amblyopic eye's central image area (i.e., the fovea), thereby forcing the visual system to use the information from the amblyopic eye's fovea. The expected treatment outcome is significant improvement in the amblyopic eye's visual acuity and in stereo vision (stereopsis).

Subjects assigned to the binocular treatment group will be prescribed the CureSight treatment to watch for ≥90 minutes per day, 5 days a week for 16 weeks for the total of <120 hours. Parents of subjects will be instructed that the 90 minutes of daily treatment should be completed in a single 90- minute session, but if this is not possible for whatever reason, the treatment may be divided into two shorter sessions totaling 90 minutes per day Subjects in the treatment group will be asked to watch digital content presented on CureSight system while wearing red/blue (anaglyph) glasses over current spectacle correction, if applicable. The subject should be instructed to sit in front of the system at the distance of ~60 cm. Positioning algorithm will automatically guide the subject to the optimal position.

Each subject will be supplied a pair of anaglyph glasses according to his/her amblyopic eye, red filter should be positioned in front of the non-amblyopic eye and the blue in front of the amblyopic eye.

In addition to the blur effect, the amblyopic eye image seen by the blue filter will have a higher intensity compared to the dominant eye red image due to the nature of the channel separation. The diameter and magnitude of the blur are adjusted during the treatment according to the VA improvement of the amblyopic eye.

In addition to the blur effect, the amblyopic eye image seen by the blue filter will have a higher intensity compared to the dominant eye red image due to the nature of the channel separation. The diameter and magnitude of the blur are adjusted during the treatment according to the VA improvement of the amblyopic eye.

Adverse Event Monitoring All adverse events which occur during the study will be reported, regardless of whether or not they are considered to be related to treatment. The following anticipated adverse events will be specifically monitored in both the therapeutic

1. Risks relating to amblyopia treatment

   * Diplopia
   * New/worsening heterotropia of greater than 10 prism diopters
   * Worsening of BCVA in either eye of 2 logMAR lines or greater from baseline
2. Risks relating to technological usage

   * Headaches
   * Eye strain
   * Skin irritation

Device deficiency Inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Including: device malfunctions, use errors, inadequate labelling of the device.

Potential device deficiencies may include:

* wrong blur position due to of eye tracker or calibration failure
* software failure
* Hardware failure; anaglyph glasses, eye tracker, computer.
* Use error such as wrong lens position, dirty lens. Risks/ Benefit discussion Standard of care treatment for amblyopia comes with the accepted risks of developing a new/worsening heterotropia or diplopia. However, the risk of developing new/worsening heterotropias or developing diplopia from the CureSight therapeutic is expected to be no greater than it would be with standard of care. In a 2016 study comparing binocular treatment to patching, the rate of new heterotropias was 8.8% in the binocular group and 5.9% in the patching group, a statistically and clinically insignificant difference. The same study showed that diplopia was rare after both treatments The procedures to be conducted in the study during visits are part of daily eye-care practice and pose no known risks. As part of a routine eye-care exam, the participant may receive cycloplegic eye drops.

The participants in both groups will be unable to perform any amblyopia treatment other than the intervention they are prescribed for the duration the study.

The diagnosis and management of reverse amblyopia is left to the investigator's judgment. Given the relatively short study duration of 16 weeks, it is believed that the risk of delaying standard of care treatment is minimal and justified.

acuity in any previous study of 2 hours of daily patching. This current proposed study is not a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* amblyopia

Exclusion Criteria:

* lack of brain and eye capacity for improved vision lack of home WiFi

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 2-6 months
  Amblyopic eye best corrected visual acuity

SECONDARY OUTCOMES:
stereopsis | 2-6 months
  depth perception- Titmus and PDI Check

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Arnold, MD, Principal Investigator — Alaska Blind Child Discovery
Locations (1):
- Alaska Blind Child Discovery, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wygnanski-Jaffe T, Kushner BJ, Moshkovitz A, Belkin M, Yehezkel O; CureSight Pivotal Trial Group. An Eye-Tracking-Based Dichoptic Home Treatment for Amblyopia: A Multicenter Randomized Clinical Trial. Ophthalmology. 2023 Mar;130(3):274-285. doi: 10.1016/j.ophtha.2022.10.020. Epub 2022 Oct 26. PMID 36306974
- [Derived] Arnold RW. Dichoptic Rescue for Spectacle-Flip Sabotage of Anisometropic Amblyopia Therapy. Clin Optom (Auckl). 2024 Mar 5;16:83-87. doi: 10.2147/OPTO.S454342. eCollection 2024. PMID 38476961